CLINICAL TRIAL: NCT02889367
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Escalation Study to Evaluate the Pharmacokinetics and the Effect on Cardiac Repolarization of Odalasvir Administered as a Tablet Formulation Under Fed Conditions in Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and the Effect on Cardiac Repolarization of Odalasvir Administered as a Single Dose Tablet Under Fed Conditions in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108163; 64294178HPC1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Healthy
MeSH Terms: interventions — odalasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (3):
- Treatment A (Experimental): Participants will receive odalasvir 100 milligram (mg) or odalasvir matching placebo once on Day 1.
  Interventions: Drug: Odalasvir 100 mg; Drug: Placebo
- Treatment B (Experimental): Participants will receive odalasvir 500 mg or odalasvir matching placebo once on Day 1.
  Interventions: Drug: Placebo; Drug: Odalasvir 500 mg
- Treatment C (Experimental): Participants will receive odalasvir (dose to be determined based on pharmacokinetic data from treatment A and B but no more than 1000 mg) or odalasvir matching placebo once on Day 1.
  Interventions: Drug: Placebo; Drug: Odalasvir (Up to maximum 1000 mg)

INTERVENTIONS:
Drug: Odalasvir 100 mg — Participants will receive odalasvir 2*50 mg tablet, orally once on Day 1.
  Arms: Treatment A
Drug: Placebo — Participants will receive odalasvir matching placebo, tablet, orally once on Day 1.
Drug: Odalasvir 500 mg — Participants will receive odalasvir 10*50 mg tablet, orally once on Day 1.
  Arms: Treatment B
Drug: Odalasvir (Up to maximum 1000 mg) — Participants will receive odalasvir to be decided up to maximum of 20*50 mg tablet, orally once on Day 1.
  Arms: Treatment C

SUMMARY:
The purpose of this study is to determine the relationship between the plasma concentrations of odalasvir and changes in the QT interval / QTc interval (QT corrected for heart rate) using exposure-response (ER) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Participant must be healthy on the basis of physical examination, medical history, and vital signs performed at screening
* Participant must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* Participant must have normal 12-lead electrocardiogram (ECG) and echocardiogram and must be healthy on the basis of clinical laboratory tests performed at screening
* Participant must be nonsmoker for at least 6 months prior to study drug administration

Exclusion Criteria:

* Participant with a history of clinically relevant heart rhythm disturbances including atrial, junctional, re-entry, and ventricular tachycardia, and heart blocks
* Participant with unusual T wave morphology (such as bifid T wave) likely to interfere with QTc measurements
* Participant with a past history of: Sick sinus syndrome, Cardiac arrhythmia (example, extrasystolic rhythms or tachycardia at rest). Isolated extrasystolic beats are not exclusionary, Risk factors associated with Torsade de Pointes (TdP) such as hypokalemia, Family history of short/long QT syndrome, Sudden unexplained death (including sudden infant death syndrome) in a first-degree relative (that is, sibling, offspring, or biological parent)
* Participant with any skin condition likely to interfere with ECG electrode placement or adhesion
* Participant with a breast implant or a history of thoracic surgery likely to cause abnormality of the electrical conduction through thoracic tissues
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 30 days or within a period less than 10 times the drug's half-life, whichever is longer, before the planned administration of study drug, or is currently enrolled in an investigational study
* Participant has a history of human immunodeficiency virus (HIV)-1 or HIV-2 infection positive, or tests positive for HIV-1 or HIV-2 at screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-03-04 (Actual); Study Completion 2017-03-04 (Actual)

PRIMARY OUTCOMES:
The Relationship Between the Plasma Concentrations of Odalasvir and Changes in the QT/QTc Interval Using Exposure-response (ER) Analysis | Baseline up to Day 4
  A linear mixed-effects model will assess the effect of dose and treatment on the change from baseline in QTc over time.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Odalasvir | 0 hour (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 30, 36, 48, 72 and 120 hours post-dose on Day 1
  Cmax is the maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of Odalasvir | 0 hour (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 30, 36, 48, 72 and 120 hours post-dose on Day 1
  AUC(0-last) is the area under the plasma concentration-time curve from time zero to the last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Odalasvir | 0 hour (pre-dose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 30, 36, 48, 72 and 120 hours post-dose on Day 1
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
PR Interval Changes and the Relationship Between the Plasma Concentrations of Odalasvir and PR Interval Changes Using ER Analysis | Baseline up to Day 4
  A linear mixed-effects model will assess the effect of dose and treatment on the change from baseline in the PR interval over time.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | up to Day 65

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States